CLINICAL TRIAL: NCT05344677
Title: Effect Of Trendelenburg Position, Warm Pad Application and Deep Breathing Exercise on Shoulder Pain and Post Gynecologic Laparoscopic Recovery
Brief Title: Shoulder Pain and Post Gynecologic Laparoscopic Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1527122021
Record Dates: First submitted 2022-03-21; First posted 2022-04-25 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-03

CONDITIONS: Gynecologic Nursing; Postoperative Pain
Keywords: Shoulder Pain after Gynecologic Laparoscopic
MeSH Terms: conditions — Pain, Postoperative | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- trendlenburg position group (Experimental): in which the women will be positioned in a Trendelenburg position (20 °) once fully awake and cooperative in the recovery room and will remain in this posture for the first 24 hrs postoperatively. The maximum time allowed in a straight-up position will be three 15-min intervals over a 24-h period
  Interventions: Other: Trendelenburg Position
- warm pad application group (Experimental): in this group warm pad (38◦C -40◦C) will be applied on the shoulder after four hours postoperatively for a period of 5-10 minutes. Each woman will be asked to place heat pads when needed during the first 24 hours.
  Interventions: Other: Warm Pad Application
- deep breathing group (Experimental): the researcher will instruct women after the end of surgery and upon consciousness to take slowly deep breathing while observing her chest and hold her breath for about 5 seconds and then exhale slowly, repeating this deep breathing technique five times after full vigilance within the first 3 hours after surgery. Then, the process will be repeated 6, 12, and 24 h later. The patient will be instructed about this type of breathing before surgery by researchers
  Interventions: Behavioral: Deep Breathing Exercise

INTERVENTIONS:
Other: Trendelenburg Position — Group 1 (trendlenburg position group) in which the women will be positioned in a Trendelenburg position (20 °) once fully awake and cooperative in the recovery room and will remain in this posture for the first 24 hrs postoperatively. The maximum time allowed in a straight-up position will be three 15-min intervals over a 24-h period.
  Arms: trendlenburg position group
Other: Warm Pad Application — • Group 2 (warm pad application group) in this group warm pad (38◦C -40◦C) will be applied on the shoulder after four hours postoperatively for a period of 5-10 minutes. Each woman will be asked to place heat pads when needed during the first 24 hours.
  Arms: warm pad application group
Behavioral: Deep Breathing Exercise — • Group 3: (deep breathing group) the researcher will instruct women after the end of surgery and upon consciousness to take slowly deep breathing while observing her chest and hold her breath for about 5 seconds and then exhale slowly, repeating this deep breathing technique five times after full vigilance within the first 3 hours after surgery. Then, the process will be repeated 6, 12, and 24 h later. The patient will be instructed about this type of breathing before surgery by researchers.
  Arms: deep breathing group

SUMMARY:
The present study aims to investigate the effect of postoperative trendelenburg position versus warm pad application and deep breathing technique on shoulder pain intensity and post gynaecologic laparoscopic recovery

DETAILED DESCRIPTION:
Laparoscopic gynecologic surgery has evolved from a limited surgical procedure used only for diagnostic purposes to a major surgical approach for treating a multitude of malignant and non-malignant pathologies. It is currently considered one of the most common surgical procedures performed by gynecologists. Laparoscopic surgery, has become widely recognized as a viable alternative to traditional laparotomy in treatment of different gynecologic diseases . The advantages of laparoscopic surgery over traditional laparotomy include a smaller surgical wound, less postoperative pain, a shorter hospital stay, faster recovery, and a better cosmetic result. However, post-laparoscopic shoulder pain (PLSP), is a prevalent complaint following laparoscopic surgery with an incidence as high as 80%. The pain can be severe and is usually relieved in 24-48h, but rarely persists for over 72h after surgery. It has also been found that PLSP is less responsive to treatment than incision and visceral pain.

The precise mechanism of post-laparoscopic shoulder pain remains unclear. Carbon dioxide accumulation and phrenic nerve irritation as a result of diaphragmatic stretching are the most accepted explanations. A number of techniques that are proposed to diminish shoulder pain as intraperitoneal instillation of local anesthetics, pulmonary recruitment maneuver, warm and humidified dioxide, low pressure pneumoperitoneum and intraperitoneal normal saline infusion. Unfortunately, these interventions have often found quite varied and sometimes even conflicting results regarding their effectiveness.

Optimal pain management is imperative for the success of immediate and long term rehabilitation. Therefore, relieving PLSP is a problem that can no longer be ignored. Effective pain control is best achieved through a combination of both pharmaceutical and non-pharmaceutical therapies. Non pharmacological methods increase women/Patient control of her feeling, improve the activity level and functional capacity and reduce dosage of analgesic drugs thus decreasing the side effects of treatment.

One of the popular non-pharmacological techniques is heat therapy, it is easy to use, inexpensive, require no prior practice, and have minimal side effects when used properly. In addition to being used for pain relief, heat is used to relieve chills or trembling, decrease joint stiffness, reduce muscle spasm, and increase connective tissue extensibility

Also, one of the recommended non-pharmacological actions is to use deep breathing relaxation techniques. The technique of breathing relaxation itself is an act of nursing care, which in this case the nurse teaches the patients how to do deep breathing techniques, slow breathing (hold inspiration to the maximum) and how to exhale slowly. In addition to reducing pain intensity, deep breathing relaxation techniques can also improve lung ventilation and increase blood oxygenation.

In addition, the trendelenburg position might decrease shoulder pain by reducing the mechanical pressure exerted by CO2 on the diaphragm and the upper abdominal muscles. CO2, known for its high solubility, would also be displaced to the pelvis that has a rich vasculature which in turn speeds up the resorption of pneumoperitoneum .However, evidence-based research is still needed in the area of pain relief after gynecologic laparoscopy and few studies have attempted to identify the effect of warm application and trendelenburg position versus deep breathing technique on PLSP. So, the purpose of this study is to determine the effect of postoperative trendelenburg position, warm application, and deep breathing exercise on shoulder pain

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-70 years
* women who were scheduled for diagnostic or operative gynecological laparoscopic surgery for non-malignant pathologies (e.g., hysterectomy, ovarian cystectomy)
* Free from any Medical history of deep vein thrombosis,shoulder surgery and chronic shoulder pain.

Exclusion Criteria:

• women with any medical or gynecological risk factors such as, morbid obese (BMI > 45) and pelvic inflammatory disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women were scheduled for diagnostic or operative gynecological laparoscopic surgery
Enrollment: 90 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NRS) | Pain intensity will be evaluated for all groups up to 24 hours postoperative
  It will be used to assess the severity of shoulder pain. Women will be instructed to choose a number from 0 to 10 that best describes their current pain.
Postoperative Quality of Recovery scale(QoR40)Postoperative Quality of Recovery scale(QoR40) | postoperative recovery will be evaluated for all groups up to 24 hours postoperative
  This tool was originally developed by Myles (2000), it is used to measure quality of recovery. It is consisted of 40 items, the items are grouped according to various aspects (dimensions) of recovery: emotional state (9items), physical comfort (12items), psychological support (7items), physical independence (5 items), and pain (7items). Subjects' response to each item will vary according to a 5 point likert scale, it was scored for positive item as "1= none of the time, 2=some of the time, 3= usually,4=most of time, and 5=all of the time.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Taha, Study Chair — Alexandria University
Locations (1):
- Noha Mohamed Mahmoud Hassan, Alexandria, Egypt

REFERENCES:
- [Background] Zhang H, Shu H, Yang L, Cao M, Zhang J, Liu K, Xiao L, Zhang X. Multiple-, but not single-, dose of parecoxib reduces shoulder pain after gynecologic laparoscopy. Int J Med Sci. 2012;9(9):757-65. doi: 10.7150/ijms.4916. Epub 2012 Oct 23. PMID 23136538
- [Background] Sutchritpongsa P, Tossamartworakul M. Pulmonary Recruitment Maneuver for Reducing Postoperative Shoulder Pain Incidence After Laparoscopic Gynecologic Surgery: A Prospective Randomized Controlled Trial. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S204. doi: 10.1016/j.jmig.2015.08.736. Epub 2015 Oct 15. No abstract available. PMID 27679045
- [Background] Zeeni C, Chamsy D, Khalil A, Abu Musa A, Al Hassanieh M, Shebbo F, Nassif J. Effect of postoperative Trendelenburg position on shoulder pain after gynecological laparoscopic procedures: a randomized clinical trial. BMC Anesthesiol. 2020 Jan 29;20(1):27. doi: 10.1186/s12871-020-0946-9. PMID 31996139

DOCUMENTS (1):
  • Study Protocol (2021-09-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT05344677/Prot_000.pdf